CLINICAL TRIAL: NCT01301495
Title: Prospective Evaluation of a New Covered Metal Stent for Malignant Lesions of the Esophagus
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: No participants enrolled for more than 1 year.
Sponsor: Weill Medical College of Cornell University (Other)
Collaborators: M.I.Tech Co., Ltd. (Unknown)
Responsible Party: Principal Investigator, Michel Kahaleh, Chief, Advanced Endoscopy, Weill Medical College of Cornell University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14989
Record Dates: First submitted 2011-02-17; First posted 2011-02-23 (Estimated); Last update posted 2015-06-03 (Estimated); Status verified 2015-06

CONDITIONS: Esophageal Cancer
Keywords: Esophageal Cancer, Malignant, Dysphagia, Esophagus, Cancer
MeSH Terms: conditions — Esophageal Neoplasms; Deglutition Disorders; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- HANAROSTENT covered Esophageal Stent (Experimental)
  Interventions: Device: HANAROSTENT TM covered Esophageal Stent

INTERVENTIONS:
Device: HANAROSTENT TM covered Esophageal Stent — HANAROSTENT covered Esophageal Stent for maintaining esophageal luminal patency in esophageal strictures caused by intrinsic and or extrinsic malignant tumors only and occlusion of concurrent esophageal fistula
  Other Names: HANAROSTENT

SUMMARY:
In this study, a newly designed and FDA approved fully covered metal stents will be used to palliate 20 patients with malignant lesion of the esophagus. Dysphagia score will be assessed before and after treatment to confirm efficacy

DETAILED DESCRIPTION:
The incidence of esophageal cancer is increasing, and despite advances in treatment, the prognosis is still very poor [1-4]. At presentation, between 50-60 % of patients have unresectable disease [5,6]. For these patients, palliation is the goal with a particular focus on the relief of dysphagia, which is the major etiology of morbidity [5,6]. Presently, Self expanding metal stent (SEMS) have become the treatment of choice for dysphagia associated with unresectable esophageal and GE junction malignancies.

In this study, a newly designed and FDA approved fully covered metal stents will be used to palliate 20 patients with malignant lesion of the esophagus. Dysphagia score will be assessed before and after treatment to confirm efficacy

The objectives are:

1. To evaluate if the newly fully covered metal stent , HANAROSTENT can provide adequate palliation of cancerous lesions of the esophagus;
2. To determine whether it is non-inferior in efficacy and safety to the esophageal stents currently available at UVa with minimal complications and improvement of symptoms

ELIGIBILITY:
Inclusion Criteria:

* Inoperable malignant obstruction of the esophageal or gastric cardia
* Malignant fistula between the esophagus ans respiratory tree
* Recurrent cancer after prior radiation

Exclusion Criteria:

* Patient unstable for endoscopic procedure
* Previous esophageal stenting
* Tumor growth within 2 cm of the upper esophageal sphincter
* Pregnant women (self reported, no pregnancy test will be done per protocol)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-11; Primary Completion 2013-11 (Actual); Study Completion 2013-11 (Actual)

PRIMARY OUTCOMES:
Palliation assessment based on Dysphagia Scores | 2 years
  To evaluate if the newly fully covered metal stent , HANAROSTENT can provide adequate palliation of cancerous lesions of the esophagus;

SECONDARY OUTCOMES:
Assessment of Complications and MD Anderson Dysphagia Score | 2-4 years
  To determine whether it is non-inferior in efficacy and safety to the esophageal stents currently available at UVa with minimal complications and improvement of symptoms

CONTACTS AND LOCATIONS:
Overall Officials: Michel Kahaleh, M.D., Principal Investigator — Weill Medical College of Cornell University
Locations (1):
- Weill Medical College of Cornell University, New York, New York, United States